CLINICAL TRIAL: NCT03022526
Title: Combined Spinal Epidural v. Epidural Labor Analgesia for Postpartum Depression Symptoms (COPE Trial): Pilot Randomized Control Trial
Brief Title: CSE v. Epidural for Postpartum Depression
Acronym: COPE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Grace Lim, MD, MS (Other)
Responsible Party: Sponsor-Investigator, Grace Lim, MD, MS, Assistant Professor of Anesthesiology, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PRO16060602
Record Dates: First submitted 2017-01-11; First posted 2017-01-16 (Estimated); Results first posted 2020-08-10 (Actual); Last update posted 2020-08-19 (Actual); Status verified 2020-08

CONDITIONS: Depression, Postpartum; Labor Pain
Keywords: Pregnant; Analgesia; Labor analgesia; Epidural; Combined spinal epidural
MeSH Terms: conditions — Depression, Postpartum; Labor Pain; Agnosia | interventions — Injections, Epidural; Bupivacaine; Fentanyl

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- CSE (Experimental): intrathecal bupivacaine 2.5mg + fentanyl 15mcg followed by infusion (PCEA): bupivacaine 0.083% with fentanyl 2mcg/mL: basal 8mL/hr, demand 8mL, 2 boluses per hour allowed, total maximum hourly allowance 24mL
  Interventions: Procedure: CSE; Drug: Bupivacaine / fentaNYL
- Epidural (Active Comparator): epidural bupivacaine 0.083% + fentanyl 2mcg/mL (8mL) followed by fentanyl 100mcg (2mL); follwed by infusion (PCEA): bupivacaine 0.083% with fentanyl 2mcg/mL: basal 8mL/hr, demand 8mL, 2 boluses per hour allowed, total maximum hourly allowance 24mL
  Interventions: Procedure: Epidural; Drug: Bupivacaine / fentaNYL

INTERVENTIONS:
Procedure: CSE
  Arms: CSE
Procedure: Epidural
  Arms: Epidural
Drug: Bupivacaine / fentaNYL

SUMMARY:
The purpose of this pilot prospective randomized control trial is to compare the initiation of labor epidural analgesia by combined spinal epidural vs. epidural for the influence on risk for postpartum depression symptoms. Investigators will randomize women to the receipt of CSE or E during labor, after measuring baseline psychological, psychosocial, and psychophysical factors related to pain and depression. The immediate research goals are to understand whether the association between labor pain and PPD is modifiable through the use of tailored anesthetic techniques.

ELIGIBILITY:
Inclusion Criteria:

* Nulliparous (no prior childbirth)
* Singleton gestation
* Third trimester
* Healthy pregnancy
* English proficiency (surveys validated in English)
* Planned vaginal delivery
* Planning to use labor epidural analgesia
* Term delivery (>/= 37.0 weeks)

Exclusion Criteria:

* Severe maternal disease
* Severe fetal disease
* Delivery not at term (delivery prior to 37.0 weeks)
* Contraindications to neuraxial anesthesia known at the time of enrollment
* Cesarean delivery WITHOUT labor
* Planning to list infant for adoption
* Did not receive epidural analgesia (either CSE or E) for labor

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 61 (Actual)
Dates: Start 2017-01; Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Magee Womens Hospital of UPMC, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Centers for Disease Control and Prevention (CDC). Prevalence of self-reported postpartum depressive symptoms--17 states, 2004-2005. MMWR Morb Mortal Wkly Rep. 2008 Apr 11;57(14):361-6. PMID 18401329
- [Background] Wisner KL, Sit DK, McShea MC, Rizzo DM, Zoretich RA, Hughes CL, Eng HF, Luther JF, Wisniewski SR, Costantino ML, Confer AL, Moses-Kolko EL, Famy CS, Hanusa BH. Onset timing, thoughts of self-harm, and diagnoses in postpartum women with screen-positive depression findings. JAMA Psychiatry. 2013 May;70(5):490-8. doi: 10.1001/jamapsychiatry.2013.87. PMID 23487258
- [Background] Logsdon MC, Wisner KL, Pinto-Foltz MD. The impact of postpartum depression on mothering. J Obstet Gynecol Neonatal Nurs. 2006 Sep-Oct;35(5):652-8. doi: 10.1111/j.1552-6909.2006.00087.x. PMID 16958723
- [Background] Ding T, Wang DX, Qu Y, Chen Q, Zhu SN. Epidural labor analgesia is associated with a decreased risk of postpartum depression: a prospective cohort study. Anesth Analg. 2014 Aug;119(2):383-392. doi: 10.1213/ANE.0000000000000107. PMID 24797120
- [Background] Robertson E, Grace S, Wallington T, Stewart DE. Antenatal risk factors for postpartum depression: a synthesis of recent literature. Gen Hosp Psychiatry. 2004 Jul-Aug;26(4):289-95. doi: 10.1016/j.genhosppsych.2004.02.006. PMID 15234824
- [Background] Righetti-Veltema M, Conne-Perreard E, Bousquet A, Manzano J. Risk factors and predictive signs of postpartum depression. J Affect Disord. 1998 Jun;49(3):167-80. doi: 10.1016/s0165-0327(97)00110-9. PMID 9629946
- [Background] O'Hara MW, Wisner KL. Perinatal mental illness: definition, description and aetiology. Best Pract Res Clin Obstet Gynaecol. 2014 Jan;28(1):3-12. doi: 10.1016/j.bpobgyn.2013.09.002. Epub 2013 Oct 7. PMID 24140480
- [Background] Chapman C. The Psychophysiology of Pain by C. Richard Chapman. In: Fishman S, Ballantyne J, Rathmell JP, editors. Bonica's Management of Pain. Fourth ed. Baltimore, MD: Lippincott Williams & Wilkins; 2010. p. 375
- [Background] Gross KH, Wells CS, Radigan-Garcia A, Dietz PM. Correlates of self-reports of being very depressed in the months after delivery: results from the Pregnancy Risk Assessment Monitoring System. Matern Child Health J. 2002 Dec;6(4):247-53. doi: 10.1023/a:1021110100339. PMID 12512766
- [Background] O'Hara M, Swain A. Rates and risk of postpartum depression-A meta-analysis. Int Rev Psychiatry. 1996;8:37-54
- [Background] Schmidt RM, Wiemann CM, Rickert VI, Smith EO. Moderate to severe depressive symptoms among adolescent mothers followed four years postpartum. J Adolesc Health. 2006 Jun;38(6):712-8. doi: 10.1016/j.jadohealth.2005.05.023. PMID 16730600
- [Background] Hirst KP, Moutier CY. Postpartum major depression. Am Fam Physician. 2010 Oct 15;82(8):926-33. PMID 20949886
- [Background] Pearlstein T, Howard M, Salisbury A, Zlotnick C. Postpartum depression. Am J Obstet Gynecol. 2009 Apr;200(4):357-64. doi: 10.1016/j.ajog.2008.11.033. PMID 19318144
- [Background] Lindahl V, Pearson JL, Colpe L. Prevalence of suicidality during pregnancy and the postpartum. Arch Womens Ment Health. 2005 Jun;8(2):77-87. doi: 10.1007/s00737-005-0080-1. Epub 2005 May 11. PMID 15883651
- [Background] Davalos DB, Yadon CA, Tregellas HC. Untreated prenatal maternal depression and the potential risks to offspring: a review. Arch Womens Ment Health. 2012 Feb;15(1):1-14. doi: 10.1007/s00737-011-0251-1. Epub 2012 Jan 4. PMID 22215285
- [Background] Murray L, Arteche A, Fearon P, Halligan S, Goodyer I, Cooper P. Maternal postnatal depression and the development of depression in offspring up to 16 years of age. J Am Acad Child Adolesc Psychiatry. 2011 May;50(5):460-70. doi: 10.1016/j.jaac.2011.02.001. Epub 2011 Apr 5. PMID 21515195
- [Background] Pearson RM, Evans J, Kounali D, Lewis G, Heron J, Ramchandani PG, O'Connor TG, Stein A. Maternal depression during pregnancy and the postnatal period: risks and possible mechanisms for offspring depression at age 18 years. JAMA Psychiatry. 2013 Dec;70(12):1312-9. doi: 10.1001/jamapsychiatry.2013.2163. PMID 24108418
- [Background] Melzack R. The myth of painless childbirth (the John J. Bonica lecture). Pain. 1984 Aug;19(4):321-337. doi: 10.1016/0304-3959(84)90079-4. No abstract available. PMID 6384895
- [Background] Boudou M, Teissedre F, Walburg V, Chabrol H. [Association between the intensity of childbirth pain and the intensity of postpartum blues]. Encephale. 2007 Oct;33(5):805-10. doi: 10.1016/j.encep.2006.10.002. French. PMID 18357852
- [Background] Eisenach JC, Pan PH, Smiley R, Lavand'homme P, Landau R, Houle TT. Severity of acute pain after childbirth, but not type of delivery, predicts persistent pain and postpartum depression. Pain. 2008 Nov 15;140(1):87-94. doi: 10.1016/j.pain.2008.07.011. Epub 2008 Sep 24. PMID 18818022
- [Background] Hiltunen P, Raudaskoski T, Ebeling H, Moilanen I. Does pain relief during delivery decrease the risk of postnatal depression? Acta Obstet Gynecol Scand. 2004 Mar;83(3):257-61. doi: 10.1111/j.0001-6349.2004.0302.x. PMID 14995921
- [Background] Vigod SN, Villegas L, Dennis CL, Ross LE. Prevalence and risk factors for postpartum depression among women with preterm and low-birth-weight infants: a systematic review. BJOG. 2010 Apr;117(5):540-50. doi: 10.1111/j.1471-0528.2009.02493.x. Epub 2010 Jan 29. PMID 20121831
- [Background] Ross LE, McQueen K, Vigod S, Dennis CL. Risk for postpartum depression associated with assisted reproductive technologies and multiple births: a systematic review. Hum Reprod Update. 2011 Jan-Feb;17(1):96-106. doi: 10.1093/humupd/dmq025. Epub 2010 Jul 6. PMID 20605900
- [Background] Howard LM, Oram S, Galley H, Trevillion K, Feder G. Domestic violence and perinatal mental disorders: a systematic review and meta-analysis. PLoS Med. 2013;10(5):e1001452. doi: 10.1371/journal.pmed.1001452. Epub 2013 May 28. PMID 23723741
- [Background] Sanger C, Iles JE, Andrew CS, Ramchandani PG. Associations between postnatal maternal depression and psychological outcomes in adolescent offspring: a systematic review. Arch Womens Ment Health. 2015 Apr;18(2):147-162. doi: 10.1007/s00737-014-0463-2. Epub 2014 Oct 2. PMID 25269760

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: We aimed to have 46 participants completing the trial, so enrolled until we hit that mark (greater than 46 enrolled due to loss to follow up).
Groups:
- Combined Spinal Epidural (CSE): intrathecal bupivacaine 2.5mg + fentanyl 15mcg followed by infusion (PCEA): bupivacaine 0.083% with fentanyl 2mcg/mL: basal 8mL/hr, demand 8mL, 2 boluses per hour allowed, total maximum hourly allowance 24mL
  CSE
  Bupivacaine / fentaNYL
- Epidural: epidural bupivacaine 0.083% + fentanyl 2mcg/mL (8mL) followed by fentanyl 100mcg (2mL); follwed by infusion (PCEA): bupivacaine 0.083% with fentanyl 2mcg/mL: basal 8mL/hr, demand 8mL, 2 boluses per hour allowed, total maximum hourly allowance 24mL
  Epidural
  Bupivacaine / fentaNYL
Period: Overall Study
Arm/Group | Combined Spinal Epidural (CSE) | Epidural
Started | 31 | 30
Completed | 21 | 25
Not Completed | 10 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Combined Spinal Epidural (CSE) | Epidural | Total
Number analyzed (Participants) | 31 | 30 | 61
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.36 (4.64) | 27.56 (6.05) | 27.46 (5.37)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 30 | 61
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2
  Not Hispanic or Latino | 31 | 28 | 59
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 3 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 6 | 11
  White | 20 | 21 | 41
  More than one race | 2 | 2 | 4
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 31 | 30 | 61

OUTCOME MEASURES:

1. Primary Outcome: Edinburgh Postnatal Depression Score (EPDS)
Description: Self-completed questionnaire, electronically completed. Scores range from 0-30, with higher score indicating higher likelihood of depressive illness. A score of 10 or greater is characterized as possible depression.
Time Frame: 6 weeks
Population: Included all participants who completed electronically administered EPDS at the 6 week timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Combined Spinal Epidural (CSE) | Epidural
Number analyzed (Participants) | 22 | 24
score on a scale | 4.23 (3.93) | 4.71 (5.82)
Statistical Analysis 1: Comparison: Combined Spinal Epidural (CSE) vs Epidural; Test type: Superiority; p = 0.7463, t-test, 2 sided

2. Secondary Outcome: Pain Score on Average (BPI - Short Form)
Description: Self-completed questionnaire, electronically completed. Pain scores range from 0 (no pain) to 10 (pain as bad as you can imagine). Participants only answered this question if answered "yes" to question: "Have you had pain other than everyday kinds of pain today?"
Time Frame: 2 days postpartum
Population: Included all participants who completed electronically administered BPI short form at at the postpartum day 2 timepoint and who reported current pain at the time of assessment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Combined Spinal Epidural (CSE) | Epidural
Number analyzed (Participants) | 14 | 16
score on a scale | 4.64 (2.13) | 4.19 (2.26)
Statistical Analysis 1: Comparison: Combined Spinal Epidural (CSE) vs Epidural; Test type: Superiority; p = 0.5764, t-test, 2 sided

3. Secondary Outcome: Pain Score on Average (BPI - Short Form)
Description: as for outcome 2
Time Frame: 6 weeks postpartum
Population: Included all participants who completed electronically administered BPI short form at at the 6 week timepoint and who reported current pain at the time of assessment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Combined Spinal Epidural (CSE) | Epidural
Number analyzed (Participants) | 5 | 1
score on a scale | 3.00 (2.35) | 4.00 (0.00)
Statistical Analysis 1: Comparison: Combined Spinal Epidural (CSE) vs Epidural; Test type: Superiority; p = 0.7169, t-test, 2 sided

4. Secondary Outcome: Pain Score on Average (BPI - Short Form)
Description: as for outcome 2
Time Frame: 3 months postpartum
Population: Included all participants who completed electronically administered BPI short form at at the 3 month timepoint and who reported current pain at the time of assessment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Combined Spinal Epidural (CSE) | Epidural
Number analyzed (Participants) | 2 | 2
score on a scale | 4.50 (2.12) | 2.00 (2.83)
Statistical Analysis 1: Comparison: Combined Spinal Epidural (CSE) vs Epidural; Test type: Superiority; p = 0.4226, t-test, 2 sided

5. Secondary Outcome: Perceived Stress (PSS)
Description: Self-completed questionnaire, electronically completed. Scores range from 0-40, with higher scores indicating higher perceived stress.
Time Frame: 2 days postpartum
Population: This population includes all participants who completed the electronically administered PSS at the postpartum day 2 timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Combined Spinal Epidural (CSE) | Epidural
Number analyzed (Participants) | 25 | 28
score on a scale | 13.08 (6.80) | 12.39 (5.55)
Statistical Analysis 1: Comparison: Combined Spinal Epidural (CSE) vs Epidural; Test type: Superiority; p = 0.6873, t-test, 2 sided

6. Secondary Outcome: Number of Participants Currently Breastfeeding at 2 Days Postpartum (Yes/No)
Description: Self-completed questionnaire, electronically completed. Results represent the percentage of each arm currently breastfeeding at this time point.
Time Frame: 2 Days Postpartum
Population: This population includes all participants who completed the electronically administered breastfeeding form at the postpartum day 2 timepoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Combined Spinal Epidural (CSE) | Epidural
Number analyzed (Participants) | 25 | 28
Participants | 22 | 18
Statistical Analysis 1: Comparison: Combined Spinal Epidural (CSE) vs Epidural; Test type: Superiority; p = 0.0452, Chi-squared

7. Secondary Outcome: Number of Participants Currently Breastfeeding at 6 Weeks Postpartum (Yes/No)
Description: as for outcome 6
Time Frame: 6 weeks postpartum
Population: This population includes all participants who completed the electronically administered breastfeeding form at the 6 week timepoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Combined Spinal Epidural (CSE) | Epidural
Number analyzed (Participants) | 20 | 24
Participants | 15 | 12
Statistical Analysis 1: Comparison: Combined Spinal Epidural (CSE) vs Epidural; Test type: Superiority; p = 0.0899, Chi-squared

8. Secondary Outcome: Number of Participants Currently Breastfeeding at 3 Months Postpartum (Yes/No)
Description: as for outcome 6
Time Frame: 3 months postpartum
Population: This population includes all participants who completed the electronically administered breastfeeding form at the 3 month timepoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Combined Spinal Epidural (CSE) | Epidural
Number analyzed (Participants) | 15 | 23
Participants | 9 | 8
Statistical Analysis 1: Comparison: Combined Spinal Epidural (CSE) vs Epidural; Test type: Superiority; p = 0.1265, Chi-squared

9. Secondary Outcome: Parent-Infant Attachment (MPAS)
Description: Self-completed questionnaire, electronically completed. Scores range from 19-95, with higher scores indicating higher attachment.
Time Frame: 6 weeks postpartum
Population: This population includes all participants who completed the electronically administered MPAS at the 6 week timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Combined Spinal Epidural (CSE) | Epidural
Number analyzed (Participants) | 22 | 24
score on a scale | 84.09 (5.48) | 87.68 (5.55)
Statistical Analysis 1: Comparison: Combined Spinal Epidural (CSE) vs Epidural; Test type: Superiority; p = 0.0328, t-test, 2 sided

10. Secondary Outcome: Parent-Infant Attachment (MPAS)
Description: as for outcome 9
Time Frame: 3 months postpartum
Population: This population includes all participants who completed the electronically administered MPAS at the 3 month timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Combined Spinal Epidural (CSE) | Epidural
Number analyzed (Participants) | 15 | 23
score on a scale | 88.08 (4.01) | 88.70 (4.78)
Statistical Analysis 1: Comparison: Combined Spinal Epidural (CSE) vs Epidural; Test type: Superiority; p = 0.6824, t-test, 2 sided

11. Secondary Outcome: Child Development (ASQ-3) Personal Social Score
Description: Self-completed questionnaire, electronically completed. Scores range from 0-60, with higher scores indicating higher personal-social development.
Time Frame: 6 weeks postpartum
Population: This population includes all participants who completed the electronically administered ASQ at the 6 week timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Combined Spinal Epidural (CSE) | Epidural
Number analyzed (Participants) | 22 | 24
score on a scale | 43.64 (11.15) | 46.04 (10.21)
Statistical Analysis 1: Comparison: Combined Spinal Epidural (CSE) vs Epidural; Test type: Superiority; p = 0.449, t-test, 2 sided

12. Secondary Outcome: Child Development (ASQ-3) Personal Social Score
Description: as for outcome 11
Time Frame: 3 months postpartum
Population: This population includes all participants who completed the electronically administered ASQ at the 3 month timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Combined Spinal Epidural (CSE) | Epidural
Number analyzed (Participants) | 15 | 23
score on a scale | 45.00 (14.85) | 47.33 (10.33)
Statistical Analysis 1: Comparison: Combined Spinal Epidural (CSE) vs Epidural; Test type: Superiority; p = 0.5996, t-test, 2 sided

13. Secondary Outcome: Parenting Self-efficacy (PMP-SE)
Description: Self-completed questionnaire, electronically completed. Scores range from 20-80, with higher scores indicating higher parenting self-efficacy.
Time Frame: 6 weeks postpartum
Population: This population includes all participants who completed the electronically administered PMP-SE at the 6 week timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Combined Spinal Epidural (CSE) | Epidural
Number analyzed (Participants) | 22 | 24
score on a scale | 71.45 (6.54) | 71.92 (5.82)
Statistical Analysis 1: Comparison: Combined Spinal Epidural (CSE) vs Epidural; Test type: Superiority; p = 0.8009, t-test, 2 sided

14. Secondary Outcome: Parenting Self-Efficacy (PMP-SE)
Description: as for outcome 13
Time Frame: 3 months postpartum
Population: This population includes all participants who completed the electronically administered PMP-SE at the 3 month timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Combined Spinal Epidural (CSE) | Epidural
Number analyzed (Participants) | 15 | 23
score on a scale | 73.20 (5.92) | 74.48 (6.47)
Statistical Analysis 1: Comparison: Combined Spinal Epidural (CSE) vs Epidural; Test type: Superiority; p = 0.5422, t-test, 2 sided

15. Secondary Outcome: Edinburgh Postnatal Depression Score (EPDS)
Description: as for outcome 1
Time Frame: 3 months
Population: This population includes all participants who completed the electronically administered EPDS at the 3 month timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Combined Spinal Epidural (CSE) | Epidural
Number analyzed (Participants) | 15 | 23
score on a scale | 3.53 (3.93) | 3.96 (3.67)
Statistical Analysis 1: Comparison: Combined Spinal Epidural (CSE) vs Epidural; Test type: Superiority; p = 0.7374, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Data on adverse events were collected during the period of subject participation (e.g., 3rd trimester until 3 months postpartum, or labor until 3 months postpartum).
Arm/Group | Combined Spinal Epidural (CSE) | Epidural
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/30
Other Adverse Events (participants affected / at risk) | 0/31 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-07-15): https://cdn.clinicaltrials.gov/large-docs/26/NCT03022526/Prot_SAP_000.pdf